CLINICAL TRIAL: NCT05261620
Title: W.I.S.E.-Wine Implementation for Surgical Recovery Enhancement
Brief Title: Wine Implementation for Surgical Recovery Enhancement
Acronym: WISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Umberto Capitanio, Head of the Kidney Tumor Research Unit, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: WISE trial
Record Dates: First submitted 2021-09-16; First posted 2022-03-02 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-06

CONDITIONS: Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SoC + WISE (Experimental): Candidates for surgery and habitual consumers of alcohol-containing beverages (7-21 alcohol-containing beverages per week) with a body mass index between 18 and 30 kg/m2. Subjects assigned to the Experimental Arm will be assigned to consume exclusively during meals one glass (around 150 ml at lunch and 150 ml at dinner) of red wine containing ethanol (˜13% EtOH v/v) with a high content of phenolic compounds (800 mg of Gallic acid equivalent).
  Interventions: Dietary Supplement: red wine
- SoC (No Intervention): Control Arm subjects adhere to diet free of any alcohol-containing beverages, as normally recommended by surgeons in their clinical practice

INTERVENTIONS:
Dietary Supplement: red wine — Subjects in the intervention arm (SoC+WISE) will be assigned to consume exclusively during meals one glass (around 150 ml at lunch and 150 ml at dinner) of red wine containing ethanol (˜13% EtOH v/v) with a high content of phenolic compounds (800 mg of Gallic acid equivalent) both for woman and men. Total polyphenolic contents and antioxidant activity (Folin-Ciocalteu method with calibration curve in gallic acid), antioxidant/radical scavenger capacity [DPPH (2,2-diphenyl-1-picrylhydrazyl) test] and phenolic profiles [HPLC (High Performance Liquid Chromatography)/DAD (diode-array detector) /ESI-MS (Electrospray Ionisation Mass Spectrometry) analysis] will be performed for wine selection for the clinical trial.
  Arms: SoC + WISE

SUMMARY:
This is a monocenter, prospective randomized clinical trial. The study aims to investigate whether moderate consumption of red wine (1 unit at lunch and 1 unit at dinner) for 30 days after surgery could improve the quality of life (QoL) and health perception status of the patient, without increasing the morbidity and the toxicity related to the surgery.

DETAILED DESCRIPTION:
Participants are randomized to receive either the standard of care (SoC - no alcohol assumption) (Control Arm) or the standard of care plus wine-controlled intake (Experimental Arm). All participants are candidates for surgery and habitual consumers of alcohol-containing beverages (7-21 alcohol-containing beverages per week) with a body mass index between 18 and 30 kg/m2.

Control Arm subjects adhere to diet free of any alcohol-containing beverages, as normally recommended by surgeons in their clinical practice.

Subjects assigned to the Experimental Arm adhere to usual diet, but were instructed to "Western prudent" dietary principles of the Lyon Diet Heart study, which is the reference in terms of cardiovascular protection, to avoid supplementation of multivitamin, minerals or probiotics, to not drink more than 2 cups of coffee, black or green tea per day and to supervise the intake of food rich in phenolic compounds through providing a list of suggested foods. Subjects will be randomly assigned to consume exclusively during meals one glass (around 150 ml at lunch and 150 ml at dinner) of red wine containing ethanol (˜13% EtOH v/v) with a high content of phenolic compounds (800 mg of Gallic acid equivalent) both for woman and men. Total polyphenolic contents and antioxidant activity (Folin-Ciocalteu method with calibration curve in gallic acid), antioxidant/radical scavenger capacity [DPPH (2,2-diphenyl-1-picrylhydrazyl) test] and phenolic profiles [HPLC (High Performance Liquid Chromatography)/DAD (diode-array detector) /ESI-MS (Electrospray Ionisation Mass Spectrometry) analysis] will be performed for wine selection for the clinical trial. The wine administered for the study purposes will be chosen from a series of wines that will be proposed by the sponsor of the study. The wine with the best polyphenolic and antioxidant properties will be chosen to be administered to the enrolled patients.

For both randomized groups, SoC plus W.I.S.E and SoC only, in order to assess participant's alcohol consumption, a trained psychologist will administer the AUDIT questionnaire specific for alcoholic drinks and a qualitative interview to patients. Frequency of intake is scheduled and each participant will be allowed to drink up to a single unit of wine at lunch and a single unit of red wine at dinner per day from the first post-operative day, during all the hospital stay, and for the next 30 days

ELIGIBILITY:
Inclusion Criteria:

* 18 years-old or older
* Candidate to surgery
* Willing to follow the protocol
* Signed informed consent

Exclusion Criteria:

* Severe Chronic Kidney Disease (eGFR<30)
* Severe liver disease (Child-Pugh B or C)
* Severe heart failure (NYHA Classes III-IV)
* body mass index lower than 18 or higher than 30 kg/m2
* Pregnant woman
* Teetotal subjects
* History of alcohol abuse evaluated through AUDIT questionnaire and qualitative interview by a psychologist
* Higher than moderate alcohol intake consumers (more than 25 g of alcohol per day for women and 40 g of alcohol per day for men)
* Type I diabetes
* Severe respiratory diseases like chronic obstructive pulmonary disease (GOLD classes III-IV)
* Neurological diseases such as Alzheimer's, Parkinson's, fibromyalgia or multiple sclerosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2025-06-12 (Actual); Study Completion 2025-06-12 (Actual)

PRIMARY OUTCOMES:
Number of participants consuming red wine after surgery showing improved health perception status assessed with the Mental Health Index (MHI) of the Short Form-36 Health Survey questionnaire | 30 days
  Health perception status measured using the Mental Health Index (MHI) of the Short Form-36 Health Survey

SECONDARY OUTCOMES:
Number of Participants consuming red wine With post-operative complications assessed with Clavien-Dindo classification | 30 days
  Rate of post-operative complications according to Clavien-Dindo classification
Number of Participants consuming red wine experiencing hospital readmissions after surgery | 30 days
  Rate of hospital readmissions from surgery
Number of male Participants consuming red wine with change in sexual perceptions after surgery using IIEF questionnaire | 30 days
  To evaluate changes in sexual perceptions after surgery using IIEF questionnaire
Number of Participants consuming red wine with a change in blood oxidative stress markers assessed using ORAC (Oxygen Radical Absorbance Capacity) tests | 30 days
  Oxidative stress will be assessed using ORAC (Oxygen Radical Absorbance Capacity) tests.

CONTACTS AND LOCATIONS:
Locations (1):
- Umberto Capitanio, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kim SJ, Kim DJ. Alcoholism and diabetes mellitus. Diabetes Metab J. 2012 Apr;36(2):108-15. doi: 10.4093/dmj.2012.36.2.108. Epub 2012 Apr 17. PMID 22540046
- [Background] Chiva-Blanch G, Arranz S, Lamuela-Raventos RM, Estruch R. Effects of wine, alcohol and polyphenols on cardiovascular disease risk factors: evidences from human studies. Alcohol Alcohol. 2013 May-Jun;48(3):270-7. doi: 10.1093/alcalc/agt007. Epub 2013 Feb 13. PMID 23408240
- [Background] Roerecke M, Rehm J. Alcohol consumption, drinking patterns, and ischemic heart disease: a narrative review of meta-analyses and a systematic review and meta-analysis of the impact of heavy drinking occasions on risk for moderate drinkers. BMC Med. 2014 Oct 21;12:182. doi: 10.1186/s12916-014-0182-6. PMID 25567363
- [Background] Schrieks IC, Heil AL, Hendriks HF, Mukamal KJ, Beulens JW. The effect of alcohol consumption on insulin sensitivity and glycemic status: a systematic review and meta-analysis of intervention studies. Diabetes Care. 2015 Apr;38(4):723-32. doi: 10.2337/dc14-1556. PMID 25805864
- [Background] Gea A, Beunza JJ, Estruch R, Sanchez-Villegas A, Salas-Salvado J, Buil-Cosiales P, Gomez-Gracia E, Covas MI, Corella D, Fiol M, Aros F, Lapetra J, Lamuela-Raventos RM, Warnberg J, Pinto X, Serra-Majem L, Martinez-Gonzalez MA; PREDIMED GROUP. Alcohol intake, wine consumption and the development of depression: the PREDIMED study. BMC Med. 2013 Aug 30;11:192. doi: 10.1186/1741-7015-11-192. PMID 23988010
- [Background] Gea A, Martinez-Gonzalez MA, Toledo E, Sanchez-Villegas A, Bes-Rastrollo M, Nunez-Cordoba JM, Sayon-Orea C, Beunza JJ. A longitudinal assessment of alcohol intake and incident depression: the SUN project. BMC Public Health. 2012 Nov 7;12:954. doi: 10.1186/1471-2458-12-954. PMID 23134690
- [Background] Rosell M, De Faire U, Hellenius ML. Low prevalence of the metabolic syndrome in wine drinkers--is it the alcohol beverage or the lifestyle? Eur J Clin Nutr. 2003 Feb;57(2):227-34. doi: 10.1038/sj.ejcn.1601548. PMID 12571653
- [Background] Scrimgeour LA, Potz BA, Elmadhun NY, Chu LM, Sellke FW. Alcohol attenuates myocardial ischemic injury. Surgery. 2017 Sep;162(3):680-687. doi: 10.1016/j.surg.2017.04.014. Epub 2017 Jun 9. PMID 28602493
- [Background] Roerecke M, Rehm J. The cardioprotective association of average alcohol consumption and ischaemic heart disease: a systematic review and meta-analysis. Addiction. 2012 Jul;107(7):1246-60. doi: 10.1111/j.1360-0443.2012.03780.x. Epub 2012 Mar 21. PMID 22229788
- [Background] Cosmi F, Di Giulio P, Masson S, Finzi A, Marfisi RM, Cosmi D, Scarano M, Tognoni G, Maggioni AP, Porcu M, Boni S, Cutrupi G, Tavazzi L, Latini R; GISSI-HF Investigators. Regular wine consumption in chronic heart failure: impact on outcomes, quality of life, and circulating biomarkers. Circ Heart Fail. 2015 May;8(3):428-37. doi: 10.1161/CIRCHEARTFAILURE.114.002091. Epub 2015 Apr 29. PMID 25925415
- [Background] Gonzalez-Rubio E, San Mauro I, Lopez-Ruiz C, Diaz-Prieto LE, Marcos A, Nova E. Relationship of moderate alcohol intake and type of beverage with health behaviors and quality of life in elderly subjects. Qual Life Res. 2016 Aug;25(8):1931-42. doi: 10.1007/s11136-016-1229-2. Epub 2016 Jan 21. PMID 26797806
- [Background] Mortensen EL, Jensen HH, Sanders SA, Reinisch JM. Better psychological functioning and higher social status may largely explain the apparent health benefits of wine: a study of wine and beer drinking in young Danish adults. Arch Intern Med. 2001 Aug 13-27;161(15):1844-8. doi: 10.1001/archinte.161.15.1844. PMID 11493125
- [Background] Hansel B, Thomas F, Pannier B, Bean K, Kontush A, Chapman MJ, Guize L, Bruckert E. Relationship between alcohol intake, health and social status and cardiovascular risk factors in the Urban Paris-Ile-de-France Cohort: is the cardioprotective action of alcohol a myth? Eur J Clin Nutr. 2010 Jun;64(6):561-8. doi: 10.1038/ejcn.2010.61. Epub 2010 May 19. PMID 20485310
- [Background] Ruidavets JB, Bataille V, Dallongeville J, Simon C, Bingham A, Amouyel P, Arveiler D, Ducimetiere P, Ferrieres J. Alcohol intake and diet in France, the prominent role of lifestyle. Eur Heart J. 2004 Jul;25(13):1153-62. doi: 10.1016/j.ehj.2003.12.022. PMID 15231374
- [Background] Mizumoto A, Ohashi S, Hirohashi K, Amanuma Y, Matsuda T, Muto M. Molecular Mechanisms of Acetaldehyde-Mediated Carcinogenesis in Squamous Epithelium. Int J Mol Sci. 2017 Sep 10;18(9):1943. doi: 10.3390/ijms18091943. PMID 28891965
- [Background] Ratna A, Mandrekar P. Alcohol and Cancer: Mechanisms and Therapies. Biomolecules. 2017 Aug 14;7(3):61. doi: 10.3390/biom7030061. PMID 28805741
- [Background] Tenta R, Fragopoulou E, Tsoukala M, Xanthopoulou M, Skyrianou M, Pratsinis H, Kletsas D. Antiproliferative Effects of Red and White Wine Extracts in PC-3 Prostate Cancer Cells. Nutr Cancer. 2017 Aug-Sep;69(6):952-961. doi: 10.1080/01635581.2017.1340489. Epub 2017 Jul 25. PMID 28742384
- [Background] Turati F, Galeone C, Rota M, Pelucchi C, Negri E, Bagnardi V, Corrao G, Boffetta P, La Vecchia C. Alcohol and liver cancer: a systematic review and meta-analysis of prospective studies. Ann Oncol. 2014 Aug;25(8):1526-35. doi: 10.1093/annonc/mdu020. Epub 2014 Mar 14. PMID 24631946
- [Background] Bagnardi V, Rota M, Botteri E, Tramacere I, Islami F, Fedirko V, Scotti L, Jenab M, Turati F, Pasquali E, Pelucchi C, Galeone C, Bellocco R, Negri E, Corrao G, Boffetta P, La Vecchia C. Alcohol consumption and site-specific cancer risk: a comprehensive dose-response meta-analysis. Br J Cancer. 2015 Feb 3;112(3):580-93. doi: 10.1038/bjc.2014.579. Epub 2014 Nov 25. PMID 25422909
- [Background] Gubner NR, Delucchi KL, Ramo DE. Associations between binge drinking frequency and tobacco use among young adults. Addict Behav. 2016 Sep;60:191-6. doi: 10.1016/j.addbeh.2016.04.019. Epub 2016 Apr 22. PMID 27156220
- [Background] Sayon-Orea C, Martinez-Gonzalez MA, Bes-Rastrollo M. Alcohol consumption and body weight: a systematic review. Nutr Rev. 2011 Aug;69(8):419-31. doi: 10.1111/j.1753-4887.2011.00403.x. PMID 21790610
- [Background] Henriksen TB, Hjollund NH, Jensen TK, Bonde JP, Andersson AM, Kolstad H, Ernst E, Giwercman A, Skakkebaek NE, Olsen J. Alcohol consumption at the time of conception and spontaneous abortion. Am J Epidemiol. 2004 Oct 1;160(7):661-7. doi: 10.1093/aje/kwh259. PMID 15383410
- [Background] Popova S, Lange S, Shield K, Mihic A, Chudley AE, Mukherjee RAS, Bekmuradov D, Rehm J. Comorbidity of fetal alcohol spectrum disorder: a systematic review and meta-analysis. Lancet. 2016 Mar 5;387(10022):978-987. doi: 10.1016/S0140-6736(15)01345-8. Epub 2016 Jan 6. PMID 26777270
- [Background] Spear LP. Effects of adolescent alcohol consumption on the brain and behaviour. Nat Rev Neurosci. 2018 Apr;19(4):197-214. doi: 10.1038/nrn.2018.10. Epub 2018 Feb 15. PMID 29467469
- [Background] Brown SA, McGue M, Maggs J, Schulenberg J, Hingson R, Swartzwelder S, Martin C, Chung T, Tapert SF, Sher K, Winters KC, Lowman C, Murphy S. A developmental perspective on alcohol and youths 16 to 20 years of age. Pediatrics. 2008 Apr;121 Suppl 4(Suppl 4):S290-310. doi: 10.1542/peds.2007-2243D. PMID 18381495
- [Background] Lau A, von Dossow V, Sander M, MacGuill M, Lanzke N, Spies C. Alcohol use disorder and perioperative immune dysfunction. Anesth Analg. 2009 Mar;108(3):916-20. doi: 10.1213/ane.0b013e318193fd89. PMID 19224804
- [Background] Imtiaz S, Shield KD, Roerecke M, Samokhvalov AV, Lonnroth K, Rehm J. Alcohol consumption as a risk factor for tuberculosis: meta-analyses and burden of disease. Eur Respir J. 2017 Jul 13;50(1):1700216. doi: 10.1183/13993003.00216-2017. Print 2017 Jul. PMID 28705945
- [Background] Rocco A, Compare D, Angrisani D, Sanduzzi Zamparelli M, Nardone G. Alcoholic disease: liver and beyond. World J Gastroenterol. 2014 Oct 28;20(40):14652-9. doi: 10.3748/wjg.v20.i40.14652. PMID 25356028
- [Background] Pelucchi C, Galeone C, Tramacere I, Bagnardi V, Negri E, Islami F, Scotti L, Bellocco R, Corrao G, Boffetta P, La Vecchia C. Alcohol drinking and bladder cancer risk: a meta-analysis. Ann Oncol. 2012 Jun;23(6):1586-93. doi: 10.1093/annonc/mdr460. Epub 2011 Oct 29. PMID 22039083
- [Background] Cao Y, Willett WC, Rimm EB, Stampfer MJ, Giovannucci EL. Light to moderate intake of alcohol, drinking patterns, and risk of cancer: results from two prospective US cohort studies. BMJ. 2015 Aug 18;351:h4238. doi: 10.1136/bmj.h4238. PMID 26286216
- [Background] Sgambato A, Ardito R, Faraglia B, Boninsegna A, Wolf FI, Cittadini A. Resveratrol, a natural phenolic compound, inhibits cell proliferation and prevents oxidative DNA damage. Mutat Res. 2001 Sep 20;496(1-2):171-80. doi: 10.1016/s1383-5718(01)00232-7. PMID 11551493
- [Background] Tonnesen H, Nielsen PR, Lauritzen JB, Moller AM. Smoking and alcohol intervention before surgery: evidence for best practice. Br J Anaesth. 2009 Mar;102(3):297-306. doi: 10.1093/bja/aen401. PMID 19218371
- [Background] Tonnesen H. Alcohol abuse and postoperative morbidity. Dan Med Bull. 2003 May;50(2):139-60. PMID 12812138
- [Background] de Lorgeril M, Salen P, Martin JL, Monjaud I, Delaye J, Mamelle N. Mediterranean diet, traditional risk factors, and the rate of cardiovascular complications after myocardial infarction: final report of the Lyon Diet Heart Study. Circulation. 1999 Feb 16;99(6):779-85. doi: 10.1161/01.cir.99.6.779. PMID 9989963
- [Background] Bohn MJ, Babor TF, Kranzler HR. The Alcohol Use Disorders Identification Test (AUDIT): validation of a screening instrument for use in medical settings. J Stud Alcohol. 1995 Jul;56(4):423-32. doi: 10.15288/jsa.1995.56.423. PMID 7674678
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Rosen R, Brown C, Heiman J, Leiblum S, Meston C, Shabsigh R, Ferguson D, D'Agostino R Jr. The Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. J Sex Marital Ther. 2000 Apr-Jun;26(2):191-208. doi: 10.1080/009262300278597. PMID 10782451
- [Background] Rosen RC, Riley A, Wagner G, Osterloh IH, Kirkpatrick J, Mishra A. The international index of erectile function (IIEF): a multidimensional scale for assessment of erectile dysfunction. Urology. 1997 Jun;49(6):822-30. doi: 10.1016/s0090-4295(97)00238-0. PMID 9187685
- [Background] Onishi T, Nishikawa K, Hasegawa Y, Yamada Y, Soga N, Arima K, Yamakado K, Hoshina A, Sugimura Y. Assessment of health-related quality of life after radiofrequency ablation or laparoscopic surgery for small renal cell carcinoma: a prospective study with medical outcomes Study 36-Item Health Survey (SF-36). Jpn J Clin Oncol. 2007 Oct;37(10):750-4. doi: 10.1093/jjco/hym107. Epub 2007 Oct 17. PMID 17942577
- [Background] Namiki S, Ishidoya S, Tochigi T, Ito A, Arai Y. Quality of life after radical prostatectomy in elderly men. Int J Urol. 2009 Oct;16(10):813-9. doi: 10.1111/j.1442-2042.2009.02371.x. Epub 2009 Aug 31. PMID 19719532
- [Background] Ficarra V, Novara G, Galfano A, Stringari C, Baldassarre R, Cavalleri S, Artibani W. Twelve-month self-reported quality of life after retropubic radical prostatectomy: a prospective study with Rand 36-Item Health Survey (Short Form-36). BJU Int. 2006 Feb;97(2):274-8. doi: 10.1111/j.1464-410X.2005.05893.x. PMID 16430628